CLINICAL TRIAL: NCT05706025
Title: Pilot Study to Evaluate Utility of EnteroTracker® as a Minimally Invasive Sampling Method to Screen for Barrett's Esophagus and Esophageal Cancer
Brief Title: Study to Evaluate EnteroTracker® as a Sampling Method to Screen for Barrett's Esophagus/Esophageal Cancer
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 22-0320.cc; BIOE (Other: University of Colorado)
Record Dates: First submitted 2022-10-05; First posted 2023-01-31 (Actual); Last update posted 2025-04-06 (Actual); Status verified 2025-04

CONDITIONS: Barrett Esophagus; Esophageal Cancer
MeSH Terms: conditions — Barrett Esophagus; Esophageal Neoplasms

STUDY DESIGN:
Intervention Model Description: The EnteroTracker® is a capsule device that includes an absorbent string.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Enterotracker (Experimental): The EnteroTracker® is a capsule device that includes an absorbent string. The trailing end of the string is taped to the cheek and the capsule is swallowed with 8-12 ounces of water. The capsule dislodges the string as it travels to the proximal small intestine. The capsule continues through the remainder of the GI tract, leaving a string in the esophagus, stomach, and duodenum. Following a 60-minute dwell time, the string is removed via the subjects' mouth and processed for analysis. Subjects will be coached to ease any potential anxieties and answer any questions. A preparatory video can be used for education if desired.
  Interventions: Device: EnteroTracker

INTERVENTIONS:
Device: EnteroTracker — The EnteroTracker® is a capsule device that includes an absorbent string.

SUMMARY:
The purpose of this study is to determine whether the EnteroTracker can obtain biomarkers that have been studied to be significant in screening BE and EAC. The current standard of care is endoscopic biopsy where the pathologist will visualize the tissue under a microscope to interpret diagnosis. Another goal of this study is to understand tolerance of the procedure so it might be used in an at-home setting.

DETAILED DESCRIPTION:
This study seeks to determine the ability of a minimally invasive capsule-string device, the EnteroTracker®, to capture biomarkers associated with Barrett's Esophagus (BE) and Esophageal Adenocarcinoma (EAC). Identification of biomarkers in samples will support development of this simple-to-use, scalable, method for early screening of EAC, a cancer that accounts for the majority of esophageal cancers in the United States. In this study, the investigators plan to capture esophageal luminal content using the EnteroTracker® from patients with confirmed BE and/or EAC (test group) and healthy adults (control group). Samples will then be analyzed for series of biomarkers associated with BE and/or EAC. The investigators will test the hypothesis that the EnteroTracker® is able to capture biomarkers of interest in subjects with BE and EAC compared to healthy controls. To address this hypothesis, the investigators propose a pilot study with the following two specific aims. Evaluate the ability and tolerability of the EnteroTracker® to capture esophageal mucosal samples in adults with BE and/or EAC as well as controls and determine the ability of the EnteroTracker®-obtained BE/EAC biomarkers to distinguish between BE and/or EAC from control subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Provision to sign and date the consent form.
2. Stated willingness to comply with all study procedures and be available for the duration of the study.
3. Be a male or female aged 45 years or older.
4. Fit in the below listed inclusion criteria

Inclusion Criteria for Test Population (BE and EAC subjects):

1. Previous diagnosis of indefinite Barrett's Esophagus (IND), non-dysplastic (ND), low grade dysplasia (LGD), high grade dysplasia (HGD), and/or esophageal adenocarcinoma (EAC)
2. Able to swallow a Tylenol sized capsule
3. Diagnostic endoscopy performed within past 3 months or able to arrive early to endoscopy for EnteroTracker® to be swallowed before endoscopy

Inclusion Criteria for Control Population (otherwise healthy adults with no evidence of BE or EAC or other esophageal cancer but with GERD) 4. Able to swallow a Tylenol sized capsule 5. 45 years of age or older

1. The majority of BE and EAC patients are age 50 years and older. Fewer than 15% of the cases are found in people younger than age 55. However current literature has suggested that there has been an increase in cases among 45-65 years old [47].

6. Apparently healthy or ≥5 years of:

1. Gastroesophageal Reflux Disease (GERD) symptoms, or
2. GERD treated with proton pump inhibitor (PPI) therapy (whether symptom control was achieved or not), or
3. Any combination of treated and untreated periods if the cumulative total is at least 5 years

Exclusion Criteria:

1. History of difficulty swallowing (dysphagia) or painful swallowing (odynophagia), including swallowing pills within 3 months of EnteroTracker® procedure
2. Inability to provide written informed consent
3. Pregnant women
4. Prior EGD during which a therapeutic procedure such as, but not limited to, ablation, cryotherapy, or endoscopic mucosal resection, was performed for the treatment of BE and/or EAC
5. Known history of esophageal varices or esophageal stricture
6. Any contraindication, as deemed in Investigator's medical judgment, to undergoing the EnteroTracker® procedure
7. Oropharyngeal cancer
8. History of esophageal or gastric surgery, with exception of uncomplicated surgical fundoplication
9. History of esophageal motility disorder
10. Currently implanted Linx device

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-05-31 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2029-03-01 (Estimated)

PRIMARY OUTCOMES:
Study Esophageal Mucosal Samples using Enterotracker Device | 2 years
  Capture esophageal mucosal samples in at least 50% of the test subjects using the EnteroTracker®.
Testing Tolerability via "Post-Procedure Tolerability Survey" | 2 years
  At least 50% of subjects describe the EnteroTracker® as "Satisfactory" from taking a "Post-Procedure Tolerability Survey".
Testing difference in Biomarkers between Control and BE/EAC patients | 2 years
  At least one biomarker differentiated between BE/EAC patients and control subjects in at least 50% of test subjects. Samples will be analyzed for various biomarkers including proteins, DNA, RNA and/or methylation of DNA.

SECONDARY OUTCOMES:
Studying DNA Collection using Enterotracker Device | 2 years
  Capture at least 1 µg of DNA from the EnteroTracker® obtained mucosal samples in at least 50% of the test subjects.
Testing Symptoms via Follow Up Adverse Event assessment call | 2 years
  No more than 50% of subjects experienced more than one of the following side effects: nausea, choking, sore throat, vomiting, or chest pain.
Testing difference in Multiple Biomarkers between Control and BE/EAC patients | 2 years
  More than one biomarker differentiated between BE/EAC patients and control subjects in at least 50% of test subjects. Samples will be analyzed for various biomarkers including proteins, DNA, RNA and/or methylation of DNA.

CONTACTS AND LOCATIONS:
Overall Officials: Sachin Wani, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado, Aurora, Colorado, United States

IPD SHARING:
Plan to Share IPD: No